CLINICAL TRIAL: NCT02539511
Title: The Effect of Brief Potent Glutamatergic Modulation on Disordered Alcohol Use
Brief Title: Glutamatergic Modulation of Disordered Alcohol Use
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Elias Dakwar, Assistant Professor of Clinical Psychiatry, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7014; R21AA023010 (NIH)
Record Dates: First submitted 2015-08-21; First posted 2015-09-03 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CI-581a+MET (Experimental): Administration of CI-581a during wk 2 at 0.71 mg/kg in the context of a 5 wk course of MET
  Interventions: Drug: CI-581a; Behavioral: Motivational Enhancement Therapy (MET)
- CI-581b+MET (Active Comparator): Administration of CI-581b during wk 2 at 0.025 mg/kg in the context of a 5 wk course of MET
  Interventions: Drug: CI-581b; Behavioral: Motivational Enhancement Therapy (MET)

INTERVENTIONS:
Drug: CI-581a
  Arms: CI-581a+MET
Drug: CI-581b
  Arms: CI-581b+MET
Behavioral: Motivational Enhancement Therapy (MET)

SUMMARY:
Alcohol use disorders remain a significant public health problem. The pharmacological facilitation of behavioral treatment represents a promising strategy for addressing disordered drinking. Alcohol use disorders are recognized to be associated with various vulnerabilities that complicate the course of treatment and that may be amenable to glutamate modulators. The purpose of this randomized, double-blind, controlled trial is to test various glutamate modulators in conjunction with motivational enhancement therapy (MET) for alcohol use disorders.

DETAILED DESCRIPTION:
Individuals diagnosed with alcohol dependence will be randomized to receive a single infusion of glutamate modulators during week 2 while engaged in a 5-week course of MET. They will meet with staff twice weekly, except for week 2 during which they will present to the clinic three times. Clinic visits include MET sessions, psychiatric monitoring, assessments, and study procedures (e.g., medication administration).

ELIGIBILITY:
Inclusion Criteria:

* Active alcohol dependence. In the case of the use of other drugs, alcohol is designated as the primary drug. At least four heavy drinking day over the past 7 days (>4 drinks a day for males, >3 drinks for females) OR minimum weekly use of 35 drinks for males and 28 for females
* Physically healthy
* No adverse reactions to study medications
* 21-69 years of age
* Capacity to consent and comply with study procedures, including sufficient proficiency in English
* Seeking to reduce or stop alcohol use

Exclusion Criteria:

* Meets criteria for current major depression, bipolar disorder, schizophrenia, any psychotic illness, including substance induced psychosis, and current substance-induced mood disorder.
* Physiological dependence on another substance requiring medical management, such as opiods or benzodiazepines, excluding caffeine, nicotine, and cannabis
* Delirium, Dementia, Amnesia, Cognitive Disorders, or Dissociative disorders. Significant dissociative symptoms
* Current suicide risk or a history of suicide attempt within the past year
* Inability to safely initiate 24 hours of abstinence from alcohol; repeated inability to initiate abstinence during the trial without incurring significant withdrawal; history of severe withdrawal phenomena over the past 6 months (e.g., withdrawal-related seizure); or self-reported inability to maintain abstinence for 24 hours without substantial distress.
* Pregnant or interested in becoming pregnant during the study period
* Any of the following cardiac conditions: clinically significant left ventricular hypertrophy, angina, clinically significant arrhythmia, or mitral valve prolapse
* Unstable physical disorders which might make participation hazardous such as end-stage AIDS, hypertension (>140/90), leukopenia, active hepatitis or other liver disease with elevated transaminase levels (< 2-3 X upper limit of normal will be considered acceptable if clotting factors are normal), renal failure, epilepsy, or untreated diabetes
* Previous history of study medication misuse or abuse, and a history of an adverse reaction/experience with prior exposure to study medications
* Recent history of significant violence (past 2 years)
* First degree relative with a psychotic disorder (bipolar disorder, schizophrenia, schizoaffective disorder, or psychosis NOS)
* obesity
* On psychotropic or other medications whose effect could be disrupted by participation in the study
* BMI > 35

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-07; Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Dakwar, MD, Principal Investigator — NYSPI/Columbia
Locations (1):
- NYSPI, New York, New York, United States

REFERENCES:
- [Derived] Dakwar E, Levin F, Hart CL, Basaraba C, Choi J, Pavlicova M, Nunes EV. A Single Ketamine Infusion Combined With Motivational Enhancement Therapy for Alcohol Use Disorder: A Randomized Midazolam-Controlled Pilot Trial. Am J Psychiatry. 2020 Feb 1;177(2):125-133. doi: 10.1176/appi.ajp.2019.19070684. Epub 2019 Dec 2. PMID 31786934

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 50 participants were enrolled in the study and from those, 40 were randomized.
Groups:
- Control Group: Midazolam+MET: 50-minute intravenous infusion of the active control midazolam (0.025 mg/kg), administered during the second week of a five week regimen of motivational enhancement therapy.
- Active Group: Ketamine+MET: 50-minute intravenous infusion of ketamine (0.71 mg/kg) administered during the second week of a five week regimen of motivational enhancement therapy.
Period: Overall Study
Arm/Group | Control Group: Midazolam+MET | Active Group: Ketamine+MET
Started | 23 | 17
Completed | 17 | 17
Not Completed | 6 | 0

BASELINE CHARACTERISTICS:
Population: 40 adults with DSM-IV alcohol dependence without significant medical or psychiatric co-morbidity.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group: Midazolam+MET | Active Group: Ketamine+MET | Total
Number analyzed (Participants) | 23 | 17 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (8.3) | 50.4 (11.3) | 53 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 7 | 21
  Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 20 | 13 | 33
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 17 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Demonstrating Alcohol Abstinence in the Control (Midazolam) Group Versus the Active (Ketamine) Group
Description: Percentage of participants demonstrating alcohol abstinence in the control (midazolam) group versus the active (ketamine) group
Time Frame: 21 days post-infusion
Population: Medically healthy, treatment-seeking adults without psychiatric comorbidity and who met DSM-IV criteria for alcohol dependence and minimum use criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Control Group: Midazolam+MET | Active Group: Ketamine+MET
Number analyzed (Participants) | 23 | 17
percentage of participants | 68.6 | 98.6

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the study period and at 6 months follow up
Groups:
- Active Group: Ketamine+MET: 50-minute intravenous infusion of ketamine (0.71 mg/kg) vs. 2) administered during the second week of a five week regimen of motivational enhancement therapy.
Arm/Group | Control Group: Midazolam+MET | Active Group: Ketamine+MET
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/17
Other Adverse Events (participants affected / at risk) | 16/23 | 16/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group: Midazolam+MET (N=23) | Active Group: Ketamine+MET (N=17)
Sedation (Nervous system disorders) | 12 | 8
Headache (Vascular disorders) | 4 | 6
Mild agitation (Psychiatric disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT02539511/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT02539511/SAP_001.pdf